CLINICAL TRIAL: NCT03616249
Title: Resistance Training Improves Sleep Profile of Elderly Sarcopenic Patients: A Randomized Trail
Brief Title: Exercise and the Sleep for the Sarcopenic Elderly
Acronym: ESSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Helton De Sa Souza, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1388065
Record Dates: First submitted 2017-05-03; First posted 2018-08-06 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Sarcopenia; Sleep; Physical Activity
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Sleep; Resistance Training

STUDY DESIGN:
Intervention Model Description: The elderly are initially distributed into two groups. Sarcopenic Group and Non-Sarcopenic Group and . 1) Training group - who will carry out the resistance training for 12 weeks or; 2) control group - who did not participate in the training in the same period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sleep quality (Experimental): To compare if elderly sartcopics present sleep losses at higher levels than non-sarcopenic elderly
  Interventions: Other: Sleep
- sleep-wake cycle. (Experimental): To compare if elderly sarcopenics present sleep-wake cycle. disorders at higher levels than non-sarcopenic elderly
  Interventions: Other: Sleep
- Exercise And Sleep quality (Active Comparator): Comparing resistance training in the sarcopenician elderly showed improvements in sleep patterns.
  Interventions: Other: Sleep; Other: Resistance Exercise
- Exercise And sleep-wake cycle. (Active Comparator): Comparing resistance training in the elderly with sarcopenia presents better sleep-wake cycle.
  Interventions: Other: Sleep; Other: Resistance Exercise

INTERVENTIONS:
Other: Sleep — Initially, all volunteers will undergo the following pre and post-intervention tests: Polysomnography; Actigraphy for 10 days; Maximum exercise test; blood collection; Physical performance evaluation; Assessment of muscle strength, assessment of body composition; And application of questionnaires.
Other: Resistance Exercise — After these procedures, the sarcophagic elderly will Resistance training, will be performed according to the latest positioning of the American College of Sports Medicine for the training of the elderly . The training will last 12 weeks, 3 times / week, with intervals of 48h between the training sessions, which will have a maximum duration of 60min. The periodization of the training will be done in a linear way, in which the volunteers will be submitted to training with 1 series of 12 to 15 repetitions at 60% of 1RM in the first week; In the second week volunteers will train at 70% of 1RM, performing 2 sets of 10 to 12 repetitions; And from the third week to the end of the training period the volunteers will train at 80% of 1RM performing 3 sets of at most 8 replicates and the intervals between sets may range from 60min to 180min. The training load will be readjusted in the 6th week of training from a new 1RM test and the training will be on the same test equipment.
  Arms: Exercise And Sleep quality; Exercise And sleep-wake cycle.

SUMMARY:
International data indicate that approximately 10% of the elderly will be affected by sarcopenia, a multifactorial syndrome that leads to the progressive and generalized loss of mass and muscular strength, leading to a decrease in quality of life, increased physical dependence, fragility, morbidity And mortality. Parallel to aging, it is well described in the literature that older people present a phase advance, which promotes alteration in the sleep-wake rhythm, as well as reduction of sleep time and quality.

In this sense, two questions need to be answered: Do sarcosis elderly present major changes in sleep-wake rhythm and in sleep parameters when compared to non-sarcopenic elderly? The improvement of sarcopenia through resistance training is also related to the improvement of the sleep-wake rhythm of the sleep parameters. In order to answer these questions, the objective of the project is to evaluate whether sarcopenic individuals present changes in the sleep-wake rhythm and sleep quality at higher levels when compared to non-sarcopenic individuals and whether the benefits of resistance training for sarcopenic individuals are related to Regulation of sleep-wake rhythm and sleep patterns.

DETAILED DESCRIPTION:
Both a World Health Organization and the Brazilian Federal Government estimate that there is an abrupt increase in the number of elderly people. Data on approximately 10% of the elderly are affected by sarcopenia, a multifactorial syndrome that leads to the progressive and generalized loss of muscle mass and muscular strength, leading to a decrease in quality of life, increased physical dependence, fragility, morbidity and mortality. Parallel to the aging, well-being in the literature that the elderly present a phase advance, which promotes the change in the sleep-wake rhythm, as well as the reduction of time and sound quality.

However, the view that a sarcophagus has a multifactorial feature sparing attention is for a possible non-sleep-wake rhythm and sleeping patterns of sarcopenic seniors at higher levels that occur in non-sarcopenic elderly. Interestingly, resistance training has often been used as a form of intervention both for the treatment of sarcopenia and for regulating the sleep-wake rhythm and to improve sleep parameters.

In this sense, two questions need to be answered: Do higher sarcopenic individuals have no sleep-wake rhythm and are there no parameters when compared to non-sarcopenic elderly? The improvement of the resistance training analysis is also related to an improvement in the sleep-wake rhythm of the sleep parameters. In order to answer these questions the objective of the project is to evaluate whether elderly sarcophages present the sleep-wake rhythm and sleep quality at higher levels when compared to non-sarcopenic elderly and the benefits of resistance training for sarcopenic individuals related to rhythm regulation Sleep-wake and sleep patterns.

Trained Non-Sarcopenic Elderly Group (GIT), Trained Elderly (GIT), Trained Elderly (GIT), Trained Elderly (ESSENCE) group; Group Elderly Controls No Sarcopenic (GC) and Elderly Group Sarcopenic Controls (GCS). The GIT and GIST groups underwent resisted training above 85% of 1 RM for 12 weeks and the GC and GCS groups will participate in lectures on lifestyle improvement every 15 days but are submitted to the training protocol. All volunteers are evaluated according to sleep objectives and subjects, as well as monitoring levels of anabolic and catabolic endocrine substances, inflammatory profile, body composition, physical and muscular performance of life before, during and after the experimental period

ELIGIBILITY:
Inclusion Criteria:

Have controlled

* blood glucose,
* blood pressure
* osteoporosis
* ability to understand and perform the physical performance test batteries
* ability to training protocol safely.

Exclusion Criteria:

* Elderly patients who are undergoing pre-treatment for sarcopenia,
* Clinically unstable,
* Present unstable angina,
* Symptomatic arrhythmia (implantable cardioverter defibrillator and pacemaker),
* Abnormal prior exertion test,
* Pulmonary arterial pressure ≥ 50 mmHg,
* Chronic obstructive pulmonary disease,
* Intermittent claudication,
* Psychiatric disorder,
* Incapacitates in understanding and performing tests and,
* Incapacitate to performing physical training safely.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Polysomnography | Pre-intervention end (12 weeks) intervention
  The full polysomnography (PSG) will be performed overnight, using a digital polysomnography equipment and using the criteria indicated by the American Academy of Sleep for sleep staging (N1, N2, and N3), REM sleep, respiratory events, awakenings and periodic movements of the lower limbs.
Pitsburgh Sleep Quality Index | Pre-intervention, 6 and 12 weeks intervention
  It is a self-applicable, easily interpreted instrument that has been extensively applied to several groups of people and collecting information on complaints about sleep, subjective quality of sleep, sleep onset latency, sleep duration, sleep efficiency, sleep disorder, use of sleeping pills and diurnal dysfunctions. Therefore, the sum of the points indicate that the higher the score the worse the quality of sleep, so when the score is less than 5 it will indicate absence of sleep disorders or a good quality of sleep, whereas if the sum is greater than 5 points the indication will be impaired sleep quality and presence of sleep disorders.
Evaluation of Sleep-Wake Cycle - Actigraphy | Pre-intervention, 6 and 12 weeks intervention
  The antidote is a multidirectional accelerometer that can be used to assess the intensity, time of physical activity, the sleep and wake time of an individual over several days for 24 hours.
  Along with the actigrated volunteers will fill in a sleep diary during the same periods of use of the actigravo. The data will be analyzed using 1-minute periods in which various sleep parameters such as total sleep time, sleep efficiency, sleep latency, and wake time may also be recorded using Actiware 5.0 software (Philips Respironics) software, from an average sensitivity threshold. To characterize the circadian rhythm profile, the data will be adjusted to the cosine transformed sine model using a least squares nonlinear regression.
Biochemical Assessments | Pre-intervention, 6 and 12 weeks intervention
  For the biochemical analysis, the fasting venous blood will be collected between 07:00 and 10:00 am using EDTA or heparin coated tubes and dried tubes with serum separator. After centrifugation for 15 minutes at 1000xg, serum and plasma will be immediately distributed in small aliquots and frozen at -80°C. After that, glucose, triglycerides, total cholesterol and fractions, total testosterone and cortisol will be analyzed from the competitive enzyme binding technique; growth hormone (GH), insulin-like growth factor 1 (IGF-1), tumor necrosis factor alpha (TNF-α), interleukin-1 receptor antagonist (IL-1ra), interleukin (IL)-6 and IL-10 by the immunoenzymatic assay method (RayBio® ELISA Kits).
Short Physical Performance Battery (SPPB) - Brazilian Version | Pre-intervention, 6 and 12 weeks interventionn
  This instrument consists of 3 tests that evaluate: the static balance standing in 3 different positions (side-by-side, semi-tandem stand, tandem stand); the walking speed to be tested using a distance of 4 meters (in a predetermined round trip) and the muscular strength of the lower limbs by means of the movement of getting up and sitting in a chair (5 consecutive and without the help of the upper limbs). All tests will be performed 3x with an interval of 2 minutes (min) between them and the best result will be considered.
Manual Grip Strength Assessment | Pre-intervention, 6 and 12 weeks intervention
  Hand grip strength will be measured by a maximal isometric test using the Jamar PC5030JI hand dynamometer (Sammons Preston, Bolingbrook, IL, USA). The dominant hand will be positioned on the dynamometer according to the recommendations proposed by the American Society of Hand Therapy . After proper positioning the volunteer can perform 3 attempts of maximum manual grip with intervals that can vary between 30 and 60 seconds (sec)
Body composition | Pre-intervention, 6 and 12 weeks intervention
  For the analysis of body composition, full body scanning was used using the dual energy X-ray absorptiometry technique (DXA; Prodigy equipped with proprietary software version 13.6, GE-Lunar, Madison, WI, USA), which was held at the Exercise Physiology Sector of the Physiology Department of UNIFESP located at the Olympic Center. Height was measured by a stadiometer fixed to the wall and body mass by a properly calibrated digital scale. After these procedures, the volunteers were placed in the supine position following the references of the scanner's collection field. At the end of the scans, the body regions (body segments) were reviewed and only then was the body composition calculated.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | Pre-intervention, 6 and 12 weeks intervention
  It is a self-administered questionnaire and refers to the chances of napping in other situations of daily life. The possibility of nap is quantified on a scale ranging from zero (0) to three (3), which 0 corresponds to no chance of snoozing and 3 the high possibility of snoozing. When the sum of points is greater than 10 it will be considered as having a high chance of having excessive daytime sleepiness while score above 16 will indicate as having severe somnolence.
Insomnia Severity Index | Pre-intervention, 6 and 12 weeks intervention
  This instruments is used for quantification of severity and for the diagnosis of insomnia based on DSM-IV, assessing recent problems in the beginning and maintenance of sleep, early awakening, interference in daytime activities, concern with sleep problems and satisfaction with their patterns

CONTACTS AND LOCATIONS:
Overall Officials: Vania D'Almeida, PhD, Study Chair — Universidade Federal de São Paulo
Locations (1):
- UNIFESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No